CLINICAL TRIAL: NCT07114588
Title: Improving Sarcopenia During Chemotherapy
Brief Title: Improving Sarcopenia in Cancer Patients Undergoing Chemotherapy With High-Protein Nutritional Supplementation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ethan Nutraceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202409133RIFE
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Early-stage Sarcopenia in Adult Cancer Patients Undergoing Chemotherapy
Keywords: Sarcopenia; Cancer; Chemotherapy; Nutritional Supplement; ETHANWELL BALANCED; Muscle Strength; BCAA; Beta-glucan; Protein Intake; Fatigue
MeSH Terms: conditions — Sarcopenia; Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplement + Elastic Band Training (Experimental)
  Interventions: Dietary Supplement: ETHANWELL BALANCED; Behavioral: Elastic Band Training
- Routine Care (Control Group) (No Intervention)

INTERVENTIONS:
Dietary Supplement: ETHANWELL BALANCED — A nutritional powder providing 250 kcal, 13.5 g protein (including 6.75 g whey protein and 2740 mg BCAAs), and 166.953 mg POLYCAN® (β-glucan) per serving. Administered 3 times daily for 8 weeks.
  Arms: Nutritional Supplement + Elastic Band Training
Behavioral: Elastic Band Training — Participants perform 5 specific resistance exercises (push up & press down, straight arm lift, seated rowing, squat, seated leg raise). Each exercise is done in 3 sets of 10 reps, 3 times per week, for 8 weeks.
  Arms: Nutritional Supplement + Elastic Band Training

SUMMARY:
This study aims to investigate whether a high-protein nutritional supplement (ETHANWELL BALANCED) can help improve muscle strength and reduce fatigue in cancer patients who are at risk of sarcopenia (age- or disease-related muscle loss) during chemotherapy. Sarcopenia is common in older adults and cancer patients and can lead to weakness, poor treatment tolerance, and reduced quality of life.

Participants aged 40 and older, receiving chemotherapy, and showing early signs of sarcopenia will be randomly assigned to two groups. The experimental group will receive nutritional education and take a high-protein nutritional drink three times per day for 8 weeks. Both groups will continue their usual medical care and perform simple resistance exercises at home.

Researchers will measure changes in grip strength, fatigue, quality of life, and nutritional status over a 12-week period. This study will help determine whether early nutrition intervention can improve treatment outcomes and quality of life for cancer patients with sarcopenia.

DETAILED DESCRIPTION:
Sarcopenia is a condition characterized by loss of muscle mass and strength, frequently observed in older adults and patients undergoing cancer treatment. It contributes to poor treatment tolerance, increased fatigue, longer hospital stays, and reduced quality of life. Early nutritional support may help reduce these complications.

This study is a prospective, randomized controlled trial investigating the effects of a high-protein oral nutritional supplement (ETHANWELL BALANCED) on muscle strength, fatigue, and quality of life in cancer patients with early-stage sarcopenia during chemotherapy. Participants will be randomly assigned to either an intervention group or a control group in a 2:1 ratio.

The intervention group will receive nutritional counseling and consume three servings of ETHANWELL BALANCED per day for 8 weeks, in addition to performing home-based resistance exercises. The control group will receive standard care and perform the same exercises. Follow-up assessments will occur at baseline and at weeks 1, 2, 4, 8, and 12.

The primary aim is to determine whether early nutritional intervention can slow the progression of sarcopenia and improve patient outcomes during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 and above.
2. Patients receiving chemotherapy or expected to undergo thoracic surgery (stage I~IV)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 and SARC-F score ≥ 4.
4. Grip strength: <28kg for males and <18kg for females.
5. Conscious and able to communicate.

Exclusion Criteria:

1. Central nervous system disorders and chronic kidney failure.
2. Mental illness or inability to cooperate.
3. Expected survival period less than 3 months.
4. Gastrointestinal dysfunction-patients who have undergone gastric resection surgery or have intestinal obstruction.
5. Heart failure-NYHA class IV.
6. Uncontrollable infection diagnosed by a physician.
7. Poorly controlled diabetes diagnosed by a physician.
8. End-stage renal disease-requiring hemodialysis or peritoneal dialysis.
9. Liver cirrhosis with severe ascites.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Improve hand grip strength (HGT) | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
  Measured using an electronic hand dynamometer. Assesses change in muscle strength over the course of 12-week intervention.

SECONDARY OUTCOMES:
Improve body weight | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
Change in Brief Fatigue Inventory - Taiwanese version (BFI-T) Score | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
  Assesses changes in cancer-related fatigue using a validated Taiwanese version of the Brief Fatigue Inventory.
Change in Quality of Life (EORTC QLQ-C30) | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
  Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Assesses patient-reported physical, emotional, and social well-being.
Change in Inflammatory Markers: IL-6, CRP, TNF-α | Baseline, Week 4, Week 12
  Blood samples are analyzed for interleukin-6, C-reactive protein, and tumor necrosis factor-alpha to evaluate systemic inflammation related to sarcopenia and nutritional status.
Change in Mid-Upper Arm Circumference (MUAC) | Baseline, Week 2, Week 4, Week 8, Week 12
  Assesses changes in muscle mass via measurement of mid-upper arm circumference using the same standardized tape throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hang Wang, PhD., Principal Investigator — Hungkuang University
Locations (1):
- National Taiwan University Hospital (NTUH), Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lim JM, Lee YJ, Cho HR, Park DC, Jung GW, Ku SK, Choi JS. Extracellular polysaccharides purified from Aureobasidium pullulans SM-2001 (Polycan) inhibit dexamethasone-induced muscle atrophy in mice. Int J Mol Med. 2018 Mar;41(3):1245-1264. doi: 10.3892/ijmm.2017.3251. Epub 2017 Nov 10. PMID 29138805
- [Result] Choi JS, Kim JW, Kim KY, Cho HR, Choi IS, Ku SK. Antiosteoporotic effects of Polycan in combination with calcium lactate-gluconate in ovariectomized rats. Exp Ther Med. 2014 Sep;8(3):957-967. doi: 10.3892/etm.2014.1793. Epub 2014 Jun 20. PMID 25120630
- [Result] Preventing effects of exopolymers purified from (EAP) supplementation and resistance exercise on muscle aging and loss in the Korean elderly: a randomized controlled trial (vol 13, pg 237, 2021). Toxicology and Environmental Health Sciences, 2021. 13(4): p. 429-429.
- [Result] Bashir KMI, Choi JS. Clinical and Physiological Perspectives of beta-Glucans: The Past, Present, and Future. Int J Mol Sci. 2017 Sep 5;18(9):1906. doi: 10.3390/ijms18091906. PMID 28872611
- [Result] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Result] Shimomura Y, Obayashi M, Murakami T, Harris RA. Regulation of branched-chain amino acid catabolism: nutritional and hormonal regulation of activity and expression of the branched-chain alpha-keto acid dehydrogenase kinase. Curr Opin Clin Nutr Metab Care. 2001 Sep;4(5):419-23. doi: 10.1097/00075197-200109000-00013. PMID 11568504
- [Result] Chou PY, Fasman GD. Structural and functional role of leucine residues in proteins. J Mol Biol. 1973 Mar 5;74(3):263-81. doi: 10.1016/0022-2836(73)90372-0. No abstract available. PMID 4692853
- [Result] Neinast M, Murashige D, Arany Z. Branched Chain Amino Acids. Annu Rev Physiol. 2019 Feb 10;81:139-164. doi: 10.1146/annurev-physiol-020518-114455. Epub 2018 Nov 28. PMID 30485760
- [Result] Martinez-Arnau FM, Fonfria-Vivas R, Buigues C, Castillo Y, Molina P, Hoogland AJ, van Doesburg F, Pruimboom L, Fernandez-Garrido J, Cauli O. Effects of Leucine Administration in Sarcopenia: A Randomized and Placebo-controlled Clinical Trial. Nutrients. 2020 Mar 27;12(4):932. doi: 10.3390/nu12040932. PMID 32230954
- [Result] Fuchs CJ, Hermans WJH, Holwerda AM, Smeets JSJ, Senden JM, van Kranenburg J, Gijsen AP, Wodzig WKHW, Schierbeek H, Verdijk LB, van Loon LJC. Branched-chain amino acid and branched-chain ketoacid ingestion increases muscle protein synthesis rates in vivo in older adults: a double-blind, randomized trial. Am J Clin Nutr. 2019 Oct 1;110(4):862-872. doi: 10.1093/ajcn/nqz120. PMID 31250889

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT07114588/Prot_SAP_000.pdf